CLINICAL TRIAL: NCT05531877
Title: Penile Implant Intraoperative Measurements Planning Chart
Acronym: PIIMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham ZAAZAA, Associate Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PIIMP Chart
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction With Diabetes Mellitus; Erectile Dysfunction Due to Arterial Disease; Erectile Dysfunction Due to Injury; Erectile Dysfunction Due to Neuropathy; Erectile Dysfunction Following Simple Prostatectomy; Erectile Dysfunction Due to Venous Disorder; Erectile Dysfunction With Type 1 Diabetes Mellitus; Erection; Incomplete; Erectile Dysfunction Due to Endocrine Disease
Keywords: Erectile Dysfunction; Penile Implant; Penile prosthesis
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: The P.I.M.P Chart will be hung on the operative room wall and penile measurements pre and post operatively recorded as the surgery progresses together with the Penile Implant size.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing Penile Implant Surgery (Experimental): All intraoperative measurements are documented in real time. Measurements recorded are as follows:
  Preoperative Pre-ICI penile length and circumference, both in relaxed and stretched states. Preoperative post-ICI penile length and circumference, both in relaxed and stretched states. Postoperative penile length and circumference. Penile implant length and girth.
  Interventions: Diagnostic Test: Penile Prosthesis Implantation

INTERVENTIONS:
Diagnostic Test: Penile Prosthesis Implantation — Penile measurement are taken preoperatively to serve as a guide to the surgeon to optimize post-operative penile size.

SUMMARY:
This is a chart of penile size measurements where penile length and width are recorded intra-operatively prior to penile prosthesis implantation to guide the surgeon to the correct and adequate post-operative penile size

DETAILED DESCRIPTION:
The chart records preoperative penile dimensions as penile length and circumference both relaxed and stretched, both in a de-tumescent and erect state, before after intra-operative injection of 1cc Prostaglandin E1 respectively, to enhance pharmacological tumescence.

The implantation of the penile implant will resume with the cavernosal sparing technique.

After the penile prosthesis has been implanted, penile length and girth will be measured and the penile implant dimensions will be recorded in the chart.

The PIMP chart will assist the surgeon in assuring he sized the penis most adequately with the implant by taking the penile dimensions ( Length and Circumference). To assure that the penis was not oversized with the implant, the post-operative penile length should not exceed the pre-operative penile tumescent stretched length.

To assure that the penis was not undersized, the postoperative penile length should not be less than the pre-operative tumescent non-stretched penile length..

The chart will also document the patients' penile dimensions pre and post operatively and could be used as an objective tool for post-operative patient counseling and reassurance about the results of the penile implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction not responding to medical treatment

Exclusion Criteria:

* Patients refusing penile prosthesis implantation as a treatment modality for their erectile dysfunction

Ages: 21 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-10-06 (Estimated)

PRIMARY OUTCOMES:
No oversizing | Intraoperative
  Post-operative Penile Length did not exceed pre-operative pharmacologically induced erect stretched length
No undersizing | Intraoperative
  Post-operative penile length not less than pre-operative pharmacologically induced erect non-stretched penile length

SECONDARY OUTCOMES:
Adequate Girth | Intraoperative
  Post operative penile circumference not less than pre-operative pharmacologically induced erect stretched circumference

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Adham ZAAZAA, Giza
  - Adham ZAAZAA, Giza, الجيزة

IPD SHARING:
Plan to Share IPD: Yes
IPD shared within 1 year of publishing upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For one year from publishing the results
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Zaazaa A, Bayerle-Eder M, Elnabarawy R, Elbitar M, Mostafa T. Penile Hemodynamic Response to Phosphodiesterase Type V Inhibitors after Cavernosal Sparing Inflatable Penile Prosthesis Implantation: A Prospective Randomized Open-Blinded End-Point (PROBE) Study. Adv Urol. 2021 Jun 28;2021:5548494. doi: 10.1155/2021/5548494. eCollection 2021. PMID 34257646
- [Background] Zaazaa A, Mostafa T. Spontaneous Penile Tumescence by Sparing Cavernous Tissue in the Course of Malleable Penile Prosthesis Implantation. J Sex Med. 2019 Mar;16(3):474-478. doi: 10.1016/j.jsxm.2019.01.012. Epub 2019 Feb 14. PMID 30773500